CLINICAL TRIAL: NCT00687921
Title: F18-Flouride PET/CT in Acute Knee Injury. A Prospective Study
Brief Title: F18-Flouride PET/CT in Acute Knee Injury
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Einat Even-Sapir MD, PhD, Dept of Nuclear Medicine. Tel Aviv Sourasky Medical Center
Other Study IDs: TASMC-08-EE-118-CTIL
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2008-06-02 (Estimated); Status verified 2008-05

CONDITIONS: Knee Injury
Keywords: Knee trauma; MRI; arthroscopy; Patients over the age of 18 who had knee trauma intent to or had MRI assessment scheduled for arthroscopy
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — not relevant
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A: patients over the age of 18 who had knee trauma, intent to or had MRI assessment and are scheduled for arthroscopy.

SUMMARY:
18F-fluoride is a positron-emitting bone-seeking agent with favorable pharmacokinetic properties. Its uptake mechanism resembles that of 99mTc-MDP. After IV administration, 18F-fluoride diffuses through the bone capillaries into the bone extracellular fluid (ECF). Its plasma clearance is more rapid than that of 99mTc-MDP and its single-passage extraction efficiency is higher. The fast blood clearance of 18F-fluoride results in a better target- to- background ratio. Bone uptake of 18F-fluoride is two-fold higher than that of 99mTc-MDP. Combining the favorable pharmacokinetic characteristics of 18F-fluoride with the high performance of PET technology, 18F-fluoride is a valuable imaging modality of the skeleton.

There are only few manuscripts on the role of static 18F-fluoride PET for detection of lesions in patients referred for non-oncologic indications The purpose of the study is to prospectively assess the added value of Fluoride PET/CT in the clinical setting of acute knee injury. The findings of Fluoride PET/CT will be correlated with those found on arthroscopy and MRI which the currently used diagnostic techniques with a high, however, not perfect diagnostic accuracy regarding the issue of bone injury which is a critical component on the long term outcome after knee injury.

DETAILED DESCRIPTION:
We intend to inject only 5mCi of Fluoride, as we already did before, thus reducing the radiation exposure to half of that of the routine Tc-MDP bone scintigraphy.

We will refer 50 patients over the age of 18 who had knee trauma, intent to or had MRI assessment and are scheduled for arthroscopy. The compartments of the injured knee will be evaluated on each of the modalities.

Exclusion criterion is pregnancy

ELIGIBILITY:
Inclusion Criteria:

* patients over the age of 18 who had knee trauma

Exclusion Criteria:

* pregnancy
* age under 18 years

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients over the age of 18 who had knee trauma, intent to or had MRI assessment and are scheduled for arthroscopy
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-03 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
we will refer patients over the age of 18 who had knee trauma, intent to or had MRI assessment and are scheduled for arthroscopy. The compartments of the injured knee will be evaluated on each of the modalities. | 6 mounth

CONTACTS AND LOCATIONS:
Overall Officials: Einat R. Even-Sapir, MD, PhD, Principal Investigator — Tel-Aviv Sourasky Medical Center